CLINICAL TRIAL: NCT07036705
Title: Optimizing an Integrated Mind and Body Treatment for Insomnia: The SLEEPS Study 2
Acronym: SLEEPS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-41821 B; R34AT012767-01 (NIH)
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Insomnia Disorder
Keywords: Passive Body Heating; Cognitive Behavioral Therapy for Insomnia; CBT-I; Insomnia Disorder; Digital Intervention; Mood Disorders; PBH
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mood Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive (1) digital cognitive behavioral therapy for insomnia (CBT-I) or (2) digital cognitive behavioral therapy and passive body heating sessions using a sauna blanket (CBT-I+PBH).
Who Masked: Outcomes Assessor
Masking Description: The clinical outcomes assessor who conducts the post-treatment clinical interviews will be masked to study randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (CBT-I) (Active Comparator): Participants will receive digital Cognitive Behavioral Therapy for Insomnia (CBT-I).
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Cognitive Behavioral Therapy for Insomnia and Passive Body Heating (CBT-I+PBH) (Experimental): Participants will receive digital Cognitive Behavioral Therapy for Insomnia (CBT-I) and Passive Body Heating (PBH) using a sauna blanket.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I); Device: Passive Body Heating (PBH)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — Cognitive behavioral therapy for insomnia (CBT-I) is a behavioral (psychotherapeutic) intervention for insomnia disorder. Participants will complete digital CBT-I online using the Sleep Healthy Using the Internet (SHUTi) program.
Device: Passive Body Heating (PBH) — Passive body heating (PBH) is a body-based treatment that participants will complete using a sauna blanket, which is similar in form factor to an adult-sized sleeping bag (head is not within the heated area). Participants will complete at least three 15-minute PBH sessions per week. Participants will complete PBH sessions in the sauna blanket placed on the floor or on a couch (i.e., not in their bed) at a setting of Level 6, 1-2 hours before bed.
  Arms: Cognitive Behavioral Therapy for Insomnia and Passive Body Heating (CBT-I+PBH)

SUMMARY:
This two-arm randomized trial will provide digital cognitive behavioral therapy for insomnia (CBT-I) to all participants and passive body heating (PBH) sessions using a sauna blanket to half of participants over a 9-week treatment period. Participants are adults aged 18 years or older with insomnia disorder.

DETAILED DESCRIPTION:
Insomnia disorder is a common and consequential mental health problem, with prevalence estimates at approximately 10%. The American College of Physicians recommends cognitive behavioral therapy for insomnia (CBT-I), an efficacious "mind" (psychological and behavioral) treatment, as the first-line treatment for adults with insomnia. Yet, about half of individuals experience residual insomnia symptoms after CBT-I. Accordingly, researchers have sought to augment CBT-I, primarily with pharmacotherapy, but many people do not want to use pharmacologic agents due to concerns about side effects and dependence. Passive-body heating (PBH), a "body" treatment, involves heating the body via hot baths or showers, infrared sauna, or other heat sources. PBH has been found to reduce the time needed to fall asleep and to improve sleep quality. PBH may improve sleep by increasing skin temperature and decreasing core body temperature, a dynamic associated with sleep onset. CBT-I and PBH thus target distinct factors that may contribute to insomnia, and the investigators hypothesize that the combination of CBT-I and PBH holds promise as a multi-component treatment for insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* Willing to use birth control if assigned female sex at birth
* Willing to receive study text messages during participation
* Location to plug sauna blanket into regular wall outlet
* Ability to lie in sauna blanket for 15 minutes
* Ability to fit in the sauna blanket
* Daily access to the internet via computer, smartphone, or tablet
* Elevated insomnia symptoms as indexed by a score of 11 or greater on the Insomnia Severity Index (ISI) at two screening timepoints
* Primary insomnia disorder (characterized by difficulty initiating sleep) as indexed by a positive diagnosis on the Structured Clinical Interview for DSM-5 Sleep Disorders (SCISD)

Exclusion Criteria:

* Night shift or swing shift worker
* Current or planned routine body heating practices (e.g., saunas, hot tubs, long baths) within 4 hours before bed that are 10 minutes or more in duration (≥2x per week)
* Pregnant or plans to become pregnant during the participation period
* Traveling internationally between screening assessment and anticipated post-intervention assessment, or during anticipated post-follow-up assessment period (~1 week)
* Other diagnosed sleep disorders or suspected sleep disorders
* Medical conditions that might increase the risk of passive body heating using an infrared sauna blanket
* Medication use that might increase the risk of passive body heating using an infrared sauna blanket
* Mental health disorder that may better explain insomnia, require priority treatment, or be exacerbated by time in bed restriction
* Medical condition that may better explain insomnia, require priority treatment, or be exacerbated by time in bed restriction
* Lifetime diagnosis of a bipolar disorder, psychosis, or other psychotic disorder
* Current (past 3 months) major depressive disorder
* Current (past 12 months) suicidality, alcohol use disorder, other substance use disorder (except mild cannabis use disorder), panic disorder, agoraphobia, social anxiety disorder, obsessive-compulsive disorder, attention-deficit/hyperactivity disorder, post-traumatic stress disorder, and eating disorders
* If using medications for mental health treatment (e.g., antidepressant medication) must have been on a stable dose for prior 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability | 9 weeks
  Proportion of participants with a score of ≥7 on the following net promoter item: "How likely would you be to recommend participating in this study to a friend or family member with insomnia?" Responses range from "Would not recommend" (0) to "Would definitely recommend" (10).

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The final IPD dataset will include self-reported demographic data, other self-reported data (e.g., subjective sleep measures, mood symptoms), and wearable-derived sleep data (wearable-derived sleep data will be shared as nightly aggregates).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months after the publication of results and unending.
Access Criteria: Data will be accessible via the Vivli platform. To access IPD arising from this project, users must complete the Vivli data request form and sign the Vivli Data Use Agreement, which limits subsequent use to the terms of the approved request and requires that users maintain data security, and refrain from any attempts to reidentify research participants or engage in any unauthorized uses of the data. In order to get access to the data, the user must submit a valid scientific question, include a statistical analysis plan, and complete all required fields on the Vivli data request form. Vivli will review the data request for completeness. Anyone who has submitted an approved data request and signed a data use agreement on Vivli will be given access to the data. Vivli will then make the data available, without cost, to users for a set period of time. Vivli will maintain storage and access of the data for as long as it maintains scientific utility.
URL: https://vivli.org

REFERENCES:
- [Background] Haghayegh S, Khoshnevis S, Smolensky MH, Diller KR, Castriotta RJ. Before-bedtime passive body heating by warm shower or bath to improve sleep: A systematic review and meta-analysis. Sleep Med Rev. 2019 Aug;46:124-135. doi: 10.1016/j.smrv.2019.04.008. Epub 2019 Apr 19. PMID 31102877
- [Background] Lee S, Oh JW, Park KM, Lee S, Lee E. Digital cognitive behavioral therapy for insomnia on depression and anxiety: a systematic review and meta-analysis. NPJ Digit Med. 2023 Mar 25;6(1):52. doi: 10.1038/s41746-023-00800-3. PMID 36966184
- See also: Research Studies Home Page to Access Online Study Screener Survey — https://www.sealab.ucsf.edu/research